CLINICAL TRIAL: NCT07075458
Title: Effectiveness Of Magic Tricks Distraction Technique In Reducing Anxiety In 3-7 Years-Old Children During Local Anesthesia Administration
Brief Title: Effectiveness Of Magic Tricks Distraction Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A0403024PP
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups:
  Magic Rope Trick group
  Magic Thumb Sleeves group
  Tell-Show-Do (TSD) group Each group will receive a different distraction technique during local anesthesia administration. The interventions will be applied in parallel, and outcomes will be compared between groups.
Masking Description: This is an open-label study; neither participants nor investigators are blinded to the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magic Rope Trick (Experimental): Children will be distracted using a magic rope trick during local anesthesia administration.
  Interventions: Behavioral: Magic Rope Trick
- Magic Thumb Sleeves (Experimental): Children will be distracted using light-up magic thumb sleeves during local anesthesia administration
  Interventions: Behavioral: Magic Thumb Sleeves
- Tell-Show-Do (TSD) (Experimental): Children will receive the conventional Tell-Show-Do behavior management technique during local anesthesia administration
  Interventions: Behavioral: Tell-Show-Do (TSD)

INTERVENTIONS:
Behavioral: Magic Rope Trick — Children will be distracted using a magic rope trick during local anesthesia administration.
  Arms: Magic Rope Trick
Behavioral: Magic Thumb Sleeves — Children will be distracted using light-up magic thumb sleeves during local anesthesia administration
  Arms: Magic Thumb Sleeves
Behavioral: Tell-Show-Do (TSD) — Children will receive the conventional Tell-Show-Do behavior management technique during local anesthesia administration
  Arms: Tell-Show-Do (TSD)

SUMMARY:
Dental anxiety among children is a significant challenge in pediatric dentistry, often hindering effective dental care. This clinical study aims to evaluate the effectiveness of two magic tricks distraction techniques (magic rope and magic thumb sleeves) in reducing dental anxiety among children aged 3-7 years during local anesthesia administration, in comparison to the conventional Tell-Show-Do (TSD) technique. Anxiety will be measured using the Raghavendra, Madhuri, and Sujata Pictorial Scale (RMS-PS) and pulse oximeter for heart rate assessment

DETAILED DESCRIPTION:
Dental anxiety in children poses a persistent challenge in pediatric dental practice, often leading to behavioral management difficulties, compromised treatment outcomes, and long-term avoidance of dental care. One of the most anxiety-inducing procedures for young patients is the administration of local anesthesia (LA), primarily due to fear of needles, unfamiliar instruments, and perceived pain. Traditional behavioral management techniques such as the Tell-Show-Do (TSD) method have been widely used to familiarize children with the dental setting and reduce procedural anxiety. However, the effectiveness of TSD during high-stress interventions like LA injections remains under debate, especially among younger children with limited cognitive development.

In response to the need for more engaging and effective behavior guidance strategies, distraction-based techniques-particularly those involving visual and interactive elements-have gained increasing interest. Among them, thaumaturgy, or the use of magic tricks, has emerged as a novel, non-pharmacological method for anxiety reduction in pediatric patients. Magic-based interventions are believed to captivate the child's attention, stimulate curiosity, and shift focus away from the source of fear, thereby promoting relaxation and behavioral cooperation.

This randomized controlled clinical trial is designed to evaluate the efficacy of two magic trick-based distraction techniques-the magic rope and magic thumb sleeves-in reducing dental anxiety in children aged 3 to 7 years, during the administration of local anesthesia. The intervention groups will be compared to a control group managed with the conventional TSD technique.

To ensure a comprehensive and objective assessment of anxiety, the study will employ a dual-modal evaluation approach:

Subjective measurement using the Raghavendra, Madhuri, and Sujata Pictorial Scale (RMS-PS), which is specifically validated for young children and uses gender-specific real-life facial photographs to help participants express their emotional states accurately.

Objective physiological measurement using pulse oximetry to monitor heart rate (HR) continuously, as HR is a well-established indicator of sympathetic nervous system activation during stress and anxiety.

All procedures will follow standardized protocols, with a dual-operator design: one clinician will administer the behavioral intervention (magic trick or TSD), while a separate clinician, blinded to the intervention group, will perform the LA injection. This design ensures methodological rigor by minimizing operator bias and isolating the effect of the behavioral technique on anxiety.

The outcomes of this study will contribute to the growing body of evidence on non-pharmacological anxiety management strategies in pediatric dentistry and may support the integration of magic-based distraction techniques as effective alternatives or adjuncts to conventional methods such as TSD.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age group of 3 to 7 years old.
* Children without any past dental treatment experience under local anesthesia.

Exclusion Criteria:

* Children with a systemic diseases.
* Children with an extreme disruptive behavior.
* Children with acute dental pain or swelling.
* Children with problems in their intellectual functions.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in dental anxiety level as measured by RMS-PS (Raghavendra, Madhuri, and Sujata Pictorial Scale) | Baseline immediately before local anesthesia administration at the same visit-periprocedural
  Dental anxiety will be assessed using the RMS-PS scale immediately before local anesthesia administration.
Change in dental anxiety level as measured by RMS-PS (Raghavendra, Madhuri, and Sujata Pictorial Scale) | Immediately after local anesthesia administration at the same visit
  Dental anxiety will be assessed using the RMS-PS scale immediately after local anesthesia administration.
heart rate using pulse oximeter | periprocedural

CONTACTS AND LOCATIONS:
Overall Officials: Nadia farrag, phd, Study Director — Mansoura University
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All the data can be shared
Supporting Information: Study Protocol
Time Frame: Data can be available forever after I complete publication
Access Criteria: internet

REFERENCES:
- [Background] Konde S, Sumaiyya S, Agarwal M, Peethambar P. "Thaumaturgy"- A Novel Behavior-shaping Technique. Int J Clin Pediatr Dent. 2020 Jul-Aug;13(4):318-321. doi: 10.5005/jp-journals-10005-1781. PMID 33149401
- See also: Int J Clin Pediatr Dent . 2024 Dec 19;17(11):1296-1301. doi: 10.5005/jp-journals-10005-2998 — https://pmc.ncbi.nlm.nih.gov/articles/PMC11703761/